CLINICAL TRIAL: NCT05696678
Title: Improving ObsQoR-11 With Continuous Wound Infusion Versus Intrathecal Morphine After Elective Cesarean Delivery: A Randomized Double-Blinded Controlled Trial Targeting Patients' Recovery and Satisfaction
Brief Title: Improving ObsQoR-11 With Continuous Wound Infusion Versus Intrathecal Morphine After Elective Cesarean Delivery
Acronym: CIVIMEC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI has permanently left the institution
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Philippe Richebe, Director of Research, Principal Investigator, Anesthesiologist, Associate Professor, MD, PhD, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-3020
Record Dates: First submitted 2022-08-23; First posted 2023-01-25 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Quality of Recovery; Anesthesia; Postoperative Pain; Cesarean Section
Keywords: ObsQoR-11
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded and controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the anesthesiologist in charge in the operating room will be aware of treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrathecal Morphine (Control Group) (Active Comparator): Spinal anesthesia with intrathecal morphine and postoperative continuous wound infusion with sterile saline.
  Interventions: Drug: Intrathecal Morphine
- Continuous Wound Infusion (Intervention Group) (Active Comparator): Spinal anesthesia without intrathecal morphine and postoperative continuous wound infusion with ropivacaine.
  Interventions: Drug: Ropivacaine 0.2%

INTERVENTIONS:
Drug: Intrathecal Morphine — Patient will receive a spinal anesthesia with a dose of 10.5 mg of bupivacaine 0.75% (1.4 ml),10 mcg of fentanyl (0.2 ml) and 100 mcg of morphine (0.2 ml) for cesarean delivery. At the end of surgery, at wound closure, a 19 Gauge 150 mm catheter will be placed under the fascia and will be linked to an elastometric pump filled with sterile saline (600 ml). A bolus of 20 ml will be administered, and an 8 ml/h infusion will be started. The catheter will be removed at 72 hours.
  Arms: Intrathecal Morphine (Control Group)
Drug: Ropivacaine 0.2% — Patient will receive a spinal anesthesia with a dose of 10.5 mg of bupivacaine 0.75% (1.4 ml),10 mcg of fentanyl (0.2 ml) and 100 mcg of morphine (0.2 ml) for cesarean delivery. At the end of surgery, at wound closure, a 19 Gauge 150 mm catheter will be placed under the fascia and will be linked to an elastometric pump filled with sterile saline (600 ml). A bolus of 20 ml will be administered, and an 8 ml/h infusion will be started. The catheter will be removed at 72 hours.
  Arms: Continuous Wound Infusion (Intervention Group)

SUMMARY:
The purpose of this prospective randomized double-blinded and controlled study is to evaluate the quality of recovery after elective cesarean delivery using the Obstetric Quality-of-Recovery-11 (ObsQoR-11) score at 24 hours between patients receiving intrathecal morphine (ITM group) compared to patients receiving a ropivacaine continuous wound infusion (CWI group).

DETAILED DESCRIPTION:
Background:

Cesarean delivery (CD) is one of the most frequently practiced surgeries in the world. Most anesthetic techniques include the use of intrathecal morphine for post-operative analgesia. While it is the gold standard, it still carries significant side effects. Recently, other analgesic options have been evaluated. Continuous anesthetic wound infusion can provide satisfactory analgesia without intrathecal morphine administration. Quality of recovery and patients' satisfaction are patients'-oriented outcomes which are now recommended as primary aim in clinical research. However, most of previous studies evaluating different post-operative analgesia management in cesarean delivery have focused primarily only on pain scores or opioid consumption, which were not always clinically relevant even if some statistical difference was reported between groups. A new scoring tool, ObsQoR-11, have recently been validated for evaluating recovery after cesarean delivery. The goal of the present study is to demonstrate an improvement in the quality of recovery after cesarean delivery as well as in patients' satisfaction when ropivacaine continuous wound infusion is used compared to the standard management with intrathecal morphine.

Hypothesis:

The investigators hypothesized that the use of ropivacaine continuous wound infusion instead of intrathecal morphine for postoperative pain management will improve the ObsQoR-11 recovery score as well as patients' satisfaction after elective cesarean delivery.

Primary objective:

To evaluate the ObsQoR-11 score at 24 hours between patients receiving intrathecal morphine (ITM group) compared to patients receiving a ropivacaine continuous wound infusion (CWI group).

Secondary objectives:

1. To evaluate the global health score of the patient (subpart of the ObsQoR-11) between ITM and CWI patients.
2. To evaluate the quality of recovery after elective cesarean delivery using the ObsQoR-11 score at 48 and 72 hours between ITM and CWI patients.
3. To evaluate the impact of the perioperative pain management on each item of ObsQoR-11 questionnaire including the quality of care the mother can provide to her child between ITM and CWI patients.
4. To evaluate pain scores at rest, at mobilization and the worst pain score as well as the opioid consumption (morphine equivalent) in the postanesthesia care unit (PACU), at 2, 4, 6, 12, 24, 48, 72 hours and 5 and 7 days after elective cesarean delivery between ITM and CWI patients.
5. To evaluate the nausea and vomiting incidence and severity during the first 24 hours after elective cesarean delivery (2, 4, 6, 12 and 24 hours) between ITM and CWI patients.
6. To evaluate the severity of the pruritus during the first 24 hours after elective cesarean delivery (2, 4, 6, 12 and 24 hours) between ITM and CWI patients.
7. To evaluate the time to first mobilization with ambulation after elective cesarean delivery between ITM and CWI patients.

Methods:

Patients scheduled for an elective cesarean delivery performed under spinal anesthesia and meeting our inclusion criteria will be fully informed about the study protocol. Interested patients will be invited to sign the informed consent form (ICF). Included patients will be invited to answer questionnaires to collect socio-demographic and medical history data (e.g. comorbidities, pregnancy details, etc…). Patients will be randomized in one of two groups by a random computer-generated number using a 1:1 randomization ratio and variable random blocks of 4 and 6.

Each patient will receive a prophylactic antacid medication consisting of 30 mL of sodium citrate 30 minutes before the surgery.

Standard monitors will be placed on the patient including a continuous pulse oximeter, continuous electrocardiography (ECG) and noninvasive blood pressure device taking blood pressure every 2.5 minutes (Dräger Perseus® A500, Drägerwerk AG & Co. KGaA, Lübeck, Germany).

Induction and anesthesia maintenance:

The anesthesia technique will be standardized. Upon arrival in the OR, spinal anesthesia will be performed in the sitting position at the lumbar level (L2-L5) with a Whitacre needle 25 Gauge (G) (BD, Mississauga ON, Canada).

The control group (ITM) will receive a dose of 10.5 mg of bupivacaine 0.75% (1.4 ml),10 mcg of fentanyl (0.2 ml) and 100 mcg of morphine (0.2 ml). The patient will then be immediately placed in the supine position (plus tilt to the left) with a phenylephrine infusion running at 0.5 mcg/kg/min (lean body weight).

The intervention group (CWI) will receive a dose of 10.5 mg of bupivacaine 0.75% (1.4 ml), 10 mcg of fentanyl (0.2 ml). The patient will then be immediately placed in the supine position (plus tilt to the left) with a phenylephrine infusion running at 0.5 mcg/kg/min (lean body weight).

Ten minutes after the spinal injection, the sensory block will be evaluated to make sure it reaches a T4 level with the ice-test. If the sensory blockade is unsatisfactory, which means the spinal anesthesia will need to be complemented with intravenous analgesics or hypnotics, then the patient will be withdrawn from the study.

A 1.5 mcg.kg-1 phenylephrine bolus (lean body weight) will be administered if the patient presents a hypotension or nausea/vomiting episode.

Hypotension will be defined as a decrease of the mean arterial blood pressure (BP) below 80% of normal baseline (pre- spinal anesthesia injection) values (as measured before intrathecal injection) for 2 consecutive BP values.

If the hypotension persists, a phenylephrine infusion will be titrated until BP reaches an adequate value. If the mean arterial blood pressure increases above 120% of normal baseline values (for 2 consecutive BP values), the phenylephrine infusion will be diminished by steps of 0.2 mcg/kg/min.

If the heart rate decreases under 50 beats/minute while the arterial pressure remains normal, a 0.2 mg IV glycopyrrolate bolus will be administered. If the heart rate decreases under 50 beats/minute while the mean arterial pressure decreases under 80% of normal values, a 5 mg IV ephedrine bolus will also be administered. At any time during the surgery, the anesthesiologist can derogate from this protocol if he deems that the security of the patient is at risk.

Prophylactic antibiotics will be administered to each patient before the incision.

Nausea and vomiting prophylaxis will consist of metoclopramide 10 mg IV after spinal anesthesia. A rescue therapy of ondansetron 4 mg IV will be administered if the patient develops nausea or vomiting despite the prophylaxis.

After umbilical cord clamping, carbetocin 100 mcg IV will be administered.

At the end of the surgery:

In the control group (ITM), at wound closure, a 19 Gauge 150 mm catheter (InfiltraLong, PAJUNK® Medical System L.P., Norcross GA, USA) will be placed under the fascia and will be linked to an elastometric pump (Baxter International Inc., Deerfield IL, USA) filled with sterile saline (600 ml). A bolus of 20 ml will be administered, and an 8 ml/h infusion (based on previous published studies) will be started. Patients will also receive 100 mg of indomethacin and 1950 mg of acetaminophen per rectum (PR) at the end of the surgery, before the transfer to PACU.

In the intervention group (CWI), at wound closure, a 19 Gauge 150 mm catheter (InfiltraLong, PAJUNK® Medical System L.P., Norcross GA, USA) will be placed under the fascia and will be linked to an elastometric pump (Baxter International Inc., Deerfield IL, USA) filled with 0.2% ropivacaine (600 ml). A bolus of 20 ml will be administered, and an 8 ml/h infusion will be started. Patients will also receive 100 mg of indomethacin and 1950 mg of acetaminophen PR at the end of the surgery.

The placement of the catheter in the fascial plane between the fascia of the transversalis muscle and the parietal peritoneum has been validated in previous studies.

Management in postanesthesia care unit:

After cesarean delivery, the patient will be transported to the postanesthesia care unit (PACU). The patient will be discharged from PACU to the ward when specific criteria are achieved (Bromage and Aldrete scores). The arriving time at PACU will be T0. From T0, all criteria of the study will be evaluated as defined.

Management in ward:

For the management of post-operative pain, all patients will benefit from the same protocol for the following 24 hours and after:

They will receive acetaminophen 975 mg Per Oral (PO) every 6 hours (regular) and naproxen 500 mg PO Bis In Die (BID) (regular) for 72 hours.

If the pain level is deemed at more than 3/10 on a Numeric Pain Rating (NRS) scale, patients will be educated to request oxycodone 5 to 7.5 mg PO every 4 hours as needed. If oxycodone is not enough or if the patient cannot tolerate medications by mouth, morphine 5 to 7.5 mg subcutaneous (SC) every 4 hours will be administered as needed. The doses of opioids needed as rescue therapy will be noted in the patients' CRF. All opioids consumed will be converted into equi-analgesic doses of PO morphine for analysis (morphine 10 mg IV or SC = hydromorphone 1.5 mg IV or SC = oxycodone 20 mg PO).

During the hospital stay, if the patient feels nauseous enough to require medical treatment ondansetron 4 mg IV every 8 hours will be administered as needed. If the nausea is persistent, metoclopramide 10 mg IV every 4 hours will be given. The dose may be repeated after 1 hour if the patient is still symptomatic. (For a maximum dosage of metoclopramide 20 mg every 4 hours). In the event both medications fail to decrease the nausea, dimenhydrinate 50 mg every 6 hours will be available as needed.

If the patient experiences pruritus that is deemed severe enough to treat, nalbuphine 2.5 mg SC every 4 hours will be administered. If the patient is not relieved after an hour, the medication will be repeated once for a maximum dosage of 5 mg SC every 4 hours. If this medication is not enough, after being reevaluated by the nursing team an hour later, the patient will receive diphenhydramine 25 mg IV, repeatable once, for a maximum dosage of 50 mg IV every 4 hours.

The patient will receive a visit from the research team or from the nursing staff at hours 2, 4, 6, 12 and 24 after the cesarean delivery. Every time, the following elements will be noted in the patients' case report form (CRF):

* Pain scores at rest, cough, mobilization (walking) on a numerical rating scale (0 to 10)
* Pruritus level and incidence graded on a scale of 0 to 3 (0 indicating no pruritus, 1 indicating mild pruritus requiring no treatment, 2 indicating moderate pruritus responsive to treatment, and 3 indicating severe pruritus unresponsive to treatment)
* Nausea and vomiting level and incidence graded on a scale of 0 to 3 (0 indicating no nausea or vomiting, 1 indicating mild nausea requiring no treatment, 2 indicating moderate nausea responsive to treatment, and 3 indicating severe nausea unresponsive to treatment and/or vomiting) After 24 hours, the following elements will also be assessed: ObsQoR-11 questionnaire and score, total PO morphine equivalent consumed, number of medication administration required for pruritus, number of medication administration required for nausea and time of the first mobilization.

Same evaluations will be done at 48 and 72 hours. The catheter will be removed under aseptic conditions at home at 72 hours by the patient after instructions given by the nursing staff.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists status I and II
* Maternal age above 18 years' old
* Elective cesarean delivery
* Spinal anesthesia
* At least 37 weeks of gestational age
* French-speaking patients (able to read and sign the consent form)

Exclusion Criteria:

* Chronic pain
* Chronic usage of any opioids
* Cardiopathy
* Unexpected difficult spinal anesthesia requiring general anesthesia or unsatisfactory sensory blockade
* Unexpected complications requiring strong hemodynamic support (transfusions, volume challenges, multiple vasopressors, inotropic drugs…) or requiring anti-hypertensive medication (including magnesium)
* Any contraindication (e.g. coagulopathy) or patient's refusal for spinal anesthesia
* Morbid obesity (BMI > 40 at the time of delivery)
* Active labour
* Emergency CD
* Fetal abnormality or prematurity (< 37 weeks of gestational age)
* Multiple gestation
* Inability to cooperate due to language or physical/mental incapacity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
ObsQoR-11 at 24 hours | 24 hours after end of surgery
  Quality of recovery after cesarean delivery using ObsQoR-11 score at 24 hours between patients receiving intrathecal morphine (ITM) compared to patients receiving a ropivacaine continuous wound infusion CWI)

SECONDARY OUTCOMES:
Global health score | 24, 48 and 72 hours after end of surgery
  Global health score of the patient (subpart of the ObsQoR-11) between ITM and CWI patients
ObsQoR-11 at 48 and 72 hours | 48 and 72 hours after end of surgery
  Quality of recovery after elective cesarean delivery using the ObsQoR-11 score at 48 and 72 hours between ITM and CWI patients
ObsQoR-11 items | 24, 48 and 72 hours after end of surgery
  Evaluate the impact of the perioperative pain management on each item of ObsQoR-11 questionnaire including the quality of care the mother can provide to her child between ITM and CWI patients
Pain scores | In postanesthesia care unit (PACU), at 2, 4, 6, 12, 24, 48, 72 hours and 5 and 7 days after the end of surgery
  Pain scores at rest, at coughing and at mobilization after elective cesarean delivery between ITM and CWI patients
Opioid consumption | In postanesthesia care unit (PACU), at 2, 4, 6, 12, 24, 48, 72 hours and 5 and 7 days after the end of surgery
  Opioid consumption (morphine equivalent) after elective cesarean delivery between ITM and CWI patients
Nausea and vomiting score | At 2, 4, 6, 12, 24 hours after the end of surgery
  Nausea and vomiting incidence and severity during the first 24 hours after elective cesarean delivery between ITM and CWI patients
Pruritus score | At 2, 4, 6, 12, 24 hours after the end of surgery
  Pruritus incidence and severity during the first 24 hours after elective cesarean delivery between ITM and CWI patients
Time to first mobilization with ambulation | During the first 24 hours after the end of surgery
  Time to first mobilization with ambulation after elective cesarean delivery between ITM and CWI patients

CONTACTS AND LOCATIONS:
Locations (1):
- CIUSSS de l'Est de l'Ile de Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No